CLINICAL TRIAL: NCT02535741
Title: Clinical Outcome Study for the Triathlon CR Total Knee
Brief Title: Clinical Outcome Study for the Triathlon Cruciate Retaining (CR) Total Knee
Acronym: TriathlonCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-S-016
Record Dates: First submitted 2015-08-21; First posted 2015-08-31 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Total Knee Arthroplasty
Keywords: Knee Replacement; Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triathlon CR Total Knee System (Other): Primary total knee replacement
  Interventions: Device: Triathlon CR Total Knee System

INTERVENTIONS:
Device: Triathlon CR Total Knee System — Primary total knee replacement

SUMMARY:
An open label, post-market, non-randomised, historical controlled, multi-centre study of the outcomes of the Triathlon Cruciate Retaining (CR) Total Knee System.

DETAILED DESCRIPTION:
An open label, post-market, non-randomised, historical controlled, multi-centre study of the outcomes of the Triathlon Cruciate Retaining (CR) Total Knee System. The primary objective of this study will be to compare the active range of motion values for the Triathlon CR Total Knee System with those of the Scorpio CR Total Knee System, a historical control group. ROM values will be measured by use of a Goniometer according to the protocol. It is expected that the Triathlon CR Total Knee System group's range of motion is not 5 degrees worse or superior to the control group's range of motion at two-years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to sign the Ethic Commission approved, study specific Informed Patient Consent Form.
2. Patients willing and able to comply with scheduled postoperative clinical and radiographic evaluations and rehabilitation.
3. Male or non-pregnant female between the ages of 21-80 years of age at the time of surgery.
4. Patients requiring a primary total knee replacement.
5. Patients with a diagnosis of osteoarthritis (OA), traumatic arthritis (TA), or avascular necrosis (AVN).
6. Patients with intact collateral ligaments.

Exclusion Criteria:

1. Patients with inflammatory arthritis.
2. Patients that are morbidly obese, body mass index (BMI) > 40.
3. Patients with a history of total / unicompartmental reconstruction of the affected joint.
4. Patients that have had a high tibial osteotomy or femoral osteotomy.
5. Patients with neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
6. Patients with a systemic or metabolic disorder leading to progressive bone deterioration.
7. Patients that are immunologically compromised, or receiving chronic steroids (>30 days duration).
8. Patients bone stock is compromised by disease or infection which cannot provide adequate support and/or fixation to the prosthesis.
9. Patients with a knee fusion to the affected joint.
10. Patients with an active or suspected latent infection in or about the knee joint.
11. Patients with a history of total joint replacement on the opposite knee within less than 1 year.
12. Patients requiring bilateral total knee replacement.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2006-10; Primary Completion 2013-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Stukenborg-Colsman, Prof., Principal Investigator — Medizinische Universität Hannover
Locations (6):
- Koge Sygehus, Køge, Roskilde, Denmark
- Hospital District of South West Finland, Turku, Westfinland, Finland
- Germany (2):
  - DRK Klinik Baden-Baden, Baden-Baden, Baden-Wurttemberg
  - Medizinische Universität Hannover, Hanover, Lower Saxony
- Spain (2):
  - Hospital Costa del Sol, Marbella, Andalusia
  - Instituto Municipal de Asistencia Sanitaria, Barcelona

REFERENCES:
- [Background] Chaudhary R, Beaupre LA, Johnston DW. Knee range of motion during the first two years after use of posterior cruciate-stabilizing or posterior cruciate-retaining total knee prostheses. A randomized clinical trial. J Bone Joint Surg Am. 2008 Dec;90(12):2579-86. doi: 10.2106/JBJS.G.00995. PMID 19047702

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient included in the study was enrolled in October 2006. 168 cases received the Triathlon CR knee system over a 56 month period in a consecutive manner in 6 centers.
Period: Overall Study
Arm/Group | Triathlon CR Total Knee System
Started | 168
Completed | 136 (Completed cases at 2 years follow-up)
Not Completed | 32
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 10
Not completed — Exclusion criteria: Bilateral implant | 4
Not completed — Missing data | 6

BASELINE CHARACTERISTICS:
Population: 168 cases have received the Triathlon CR total knee replacement
Groups:
- Triathlon CR Total Knee System: Progressive data: Primary total knee replacement
Arm/Group | Triathlon CR Total Knee System
Number analyzed (Participants) | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114
  Male | 54
Range of Motion (ROM) [Mean (Standard Deviation); unit: degree] | 107.21 (12.5)

OUTCOME MEASURES:

1. Primary Outcome: Mean Triathlon CR Active Range of Motion (ROM)
Description: Comparison of the active ROM values for patients receiving the Triathlon CR Total Knee System with historical active ROM values of the Scorpio CR Total Knee System, a control group by literature review at 2 years post Total Knee Arthroplasty. See Chaudhary R, et al 2008 JBJS included for historical control data.
Time Frame: 2 years follow-up
Population: Comparison to data from the literature was not done.
Measure: Mean (Standard Deviation); unit: degree
Groups:
- Triathlon CR Total Knee System: Prospective data of the Triathlon CR primary total knee replacement
Arm/Group | Triathlon CR Total Knee System
Number analyzed (Participants) | 134
degree | 112.96 (13.708)

2. Secondary Outcome: Investigation of Patient Outcome With Radiographic Analysis
Description: Plain radiographs will be obtained for assessment of fixation of the device.
Time Frame: Pre-operative, 3 months, 1, 2 and 5 years follow-up
Population: Radiographic data were not collected
Arm/Group | Triathlon CR Total Knee System
Number analyzed (Participants) | 0

3. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Knee Society Score (KSS)
Description: The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, Range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: Pre-operative, 3 months, 1, 2, 3, 4 and 5 years follow-up
Population: The number included in the analysis in one or more rows differs from the overall number analysed because that data were not collected.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon CR Total Knee System
Number analyzed (Participants) | 164
units on a scale
  KSS Pain/Motion pre-operative | 38.2 (21.7)
  KSS Pain/Motion 3 months: number analyzed (Participants) | 163
  KSS Pain/Motion 3 months | 75.2 (15.4)
  KSS Pain/Motion 1 year: number analyzed (Participants) | 150
  KSS Pain/Motion 1 year | 81.7 (13.8)
  KSS Pain/Motion 2 years: number analyzed (Participants) | 131
  KSS Pain/Motion 2 years | 86 (11.5)
  KSS Pain/Motion 5 years: number analyzed (Participants) | 86
  KSS Pain/Motion 5 years | 88 (9.7)
  KSS Function Score pre-operative | 58.9 (14.2)
  KSS Function Score 3 months: number analyzed (Participants) | 159
  KSS Function Score 3 months | 78.9 (17.5)
  KSS Function Score 1 year: number analyzed (Participants) | 148
  KSS Function Score 1 year | 82.2 (18.5)
  KSS Function Score 2 years: number analyzed (Participants) | 131
  KSS Function Score 2 years | 86.2 (18)
  KSS Function Score 5 years: number analyzed (Participants) | 86
  KSS Function Score 5 years | 81.5 (20.5)

4. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Short Form 12 (SF-12) Patient Questionnaire
Description: The SF-12 Health Survey is a 12-item patient completed questionnaire to measure general health and well-being. It includes a physical (PSC) and mental status component (MCS) score; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: Pre-operative, 3 months, 1, 2, 3, 4 and 5 years follow-up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon CR Total Knee System
Number analyzed (Participants) | 163
units on a scale
  pre-operative PCS | 30.0 (8.2)
  3 months PCS: number analyzed (Participants) | 155
  3 months PCS | 37.5 (8.8)
  1 year PCS: number analyzed (Participants) | 139
  1 year PCS | 42.0 (9.4)
  2 years PCS: number analyzed (Participants) | 127
  2 years PCS | 44.6 (9.7)
  3 years PCS: number analyzed (Participants) | 125
  3 years PCS | 41.9 (10.8)
  4 years PCS: number analyzed (Participants) | 104
  4 years PCS | 42.1 (10.7)
  5 years PCS: number analyzed (Participants) | 82
  5 years PCS | 43.0 (11.1)
  pre-operative MCS | 47.5 (13.5)
  3 months MCS: number analyzed (Participants) | 154
  3 months MCS | 50.7 (10.8)
  1 year MCS: number analyzed (Participants) | 139
  1 year MCS | 52.2 (9.5)
  2 years MCS: number analyzed (Participants) | 127
  2 years MCS | 50.8 (10.5)
  3 years MCS: number analyzed (Participants) | 125
  3 years MCS | 51.4 (11.3)
  4 years MCS: number analyzed (Participants) | 104
  4 years MCS | 50.7 (10.5)
  5 years MCS: number analyzed (Participants) | 82
  5 years MCS | 53.9 (10.3)

5. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Western Ontario McMaster Osteoarthritis Index (WOMAC) Patient Questionnaire
Description: The WOMAC collects information specific to osteoarthritis outcomes. The questionnaire uses a visual analog scale for pain, measuring factors of general pain, stiffness, and physical findings. Pain is scored from 0 to 100 for each set of factors, with 0 indicating no pain and 100 indicating extreme pain. Total WOMAC scores range from 0 to 300. Lower values represent better outcomes.
Time Frame: Pre-operative, 3 months, 1, 2, 3, 4 and 5 years follow-up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon CR Total Knee System
Number analyzed (Participants) | 159
units on a scale
  pre-operative total score | 166.42 (60.88)
  3 months total score: number analyzed (Participants) | 143
  3 months total score | 78.99 (58.98)
  1 year total score: number analyzed (Participants) | 135
  1 year total score | 45.04 (47.14)
  2 years total score: number analyzed (Participants) | 122
  2 years total score | 40.6 (41.30)
  3 years total score: number analyzed (Participants) | 117
  3 years total score | 46.28 (51.02)
  4 years total score: number analyzed (Participants) | 99
  4 years total score | 47.94 (52.21)
  5 years total score: number analyzed (Participants) | 80
  5 years total score | 43.64 (53.1)

ADVERSE EVENTS:
Time Frame: 3 months, 1 year, 2 years, 5 years
Description: Adverse event data were collected for the Triathlon CR arm during the follow-up visits.
Groups:
- Triathlon CR Total Knee System: Triathlon CR Primary total knee replacement
Arm/Group | Triathlon CR Total Knee System
Serious Adverse Events (participants affected / at risk) | 23/168
Other Adverse Events (participants affected / at risk) | 0/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triathlon CR Total Knee System (N=168)
Apoplex (Nervous system disorders) | 1 (1)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 6 (6)
Loosening of tibial component (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Contralateral knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Contralateral total knee replacement (Musculoskeletal and connective tissue disorders) | 7 (7)
Hip Replacement (Musculoskeletal and connective tissue disorders) | 2 (2)
Deep joint infection (Renal and urinary disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1)
Knee instability (Musculoskeletal and connective tissue disorders) | 2 (2)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee pain, poor ROM (Vascular disorders) | 1 (1)
Multinodular goiter (Endocrine disorders) | 1 (1)
Patellar Subluxation (Musculoskeletal and connective tissue disorders) | 2 (2)
Poor ROM (Musculoskeletal and connective tissue disorders) | 1 (1)
Pulmonal infection (Infections and infestations) | 1 (1)
Soft tissue trauma (Injury, poisoning and procedural complications) | 2 (2)
Flexion Contracture (Musculoskeletal and connective tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less